CLINICAL TRIAL: NCT03341793
Title: Impact of Changes in Muscle Secretome in the Remission of Type 2 Diabetes Mellitus Induced by Bariatric Surgery
Acronym: MYDIASECRET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017/24AOU/417
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscle secretion (Experimental): Characterize the changes in muscle secretion induced by bariatric surgery and determine their role in improving the insulin sensitivity of skeletal muscle and insulin secretion by B cell responsible for the remission of diabetes mellitus.
  Interventions: Diagnostic Test: Muscle biopsy and blood test

INTERVENTIONS:
Diagnostic Test: Muscle biopsy and blood test — Characterize the changes in muscle secretion induced by bariatric surgery and determine their role in improving the insulin sensitivity of skeletal muscle and insulin secretion by B cell responsible for the remission of diabetes mellitus.

SUMMARY:
Bariatric surgery is recognized as a therapeutic modality of type 2 diabetes. The mechanisms of this remission of diabetes remain poorly understood.

The aim of our research is to characterize the changes in muscle secretome induced by bariatric surgery and to determine their role in improving the insulin sensitivity of skeletal muscle and insulin secretion by the B cell responsible for the remission of diabetes.

DETAILED DESCRIPTION:
Bariatric surgery is recognized as a therapeutic modality of type 2 diabetes. The mechanisms of this remission of diabetes remain poorly understood.

The aim of our research is to characterize the changes in muscle secretome induced by bariatric surgery and to determine their role in improving the insulin sensitivity of skeletal muscle and insulin secretion by the B cell responsible for the remission of diabetes.

This prospective study will be carried out in insulin-resistant diabetic patients or not in whom blood and muscle samples will be carried out before and after bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* Age from 19 to 69 year-old Candidate for bariatric surgery BMI ≥ 35kg / m² with at least one subsequent comorbidity (SAS or type 2 diabetes mellitus or refractory HTA) or BMI ≥ 40kg / m² Non-diabetic or diabetic with HbA1c <7.5% without treatment except metformin Caucasian No pregnancy or breastfeeding No history of neoplasia in the last 5 years No history of uncontrolled endocrinopathy other than diabetes Informed consent signed by patient

Exclusion Criteria:

* Non-caucasian Major Depression Hemorrhagic risk (biopsy) associated with taking anticoagulants/antiaggregants Known myopathy Systemic administration of steroids (> 1mg/kg in hydrocortisone) Hyperthyroidism Type 1 diabetes Psychological, familial, sociological or geographical condition potentially limiting compliance with the protocol Participation in other clinical drug studies Modification of anti-diabetic treatment during the month preceding surgery

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in myokine (muscle secretome) secretion induced by bariatric surgery | Level of myokines in culture media conditioned by muscle cells taken before and 3 months after bariatric surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
There no plan at this moment

REFERENCES:
- [Derived] Orioli L, Canouil M, Sawadogo K, Ning L, Deldicque L, Lause P, de Barsy M, Froguel P, Loumaye A, Deswysen Y, Navez B, Bonnefond A, Thissen JP. Identification of myokines susceptible to improve glucose homeostasis after bariatric surgery. Eur J Endocrinol. 2023 Sep 1;189(3):409-421. doi: 10.1093/ejendo/lvad122. PMID 37638789